CLINICAL TRIAL: NCT06203574
Title: Clinical Study of TROP-2 PET/CT for Noninvasive Diagnosis of Solid Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, YiHui Guan, Professor, Huashan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KY2023-1017
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Positron-Emission Tomography; Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with solid tumors (Experimental): Subjects were recruited from Huashan Hospital of Fudan University.
  Interventions: Radiation: [68Ga]Ga-NOTA-T4 or [18F]AlF-RESCA-T4

INTERVENTIONS:
Radiation: [68Ga]Ga-NOTA-T4 or [18F]AlF-RESCA-T4 — The dose of [68Ga]Ga-NOTA-T4 or [18F]AlF-RESCA-T4 was calculated based on the patient's body weight to be 3.7 MBq [0.1 mCi]/kg, and the method of administration was intravenous push, with one single imaging administration.

SUMMARY:
This study will investigate the safety and preliminary diagnostic efficacy of [68Ga]Ga-NOTA-T4 or [18F]AlF-RESCA-T4 in pancreatic cancer, breast cancer, head and neck cancer, lung cancers and other types of solid tumors. Then, this study will provide a new method for the noninvasive target-specific diagnosis of pancreatic cancer, breast cancer, head and neck cancer, lung cancers and other types of solid tumors. PET imaging of TROP-2 will be integrated to TROP-2-targeted therapies in some of the included patients. Therefore, PET imaging with [68Ga]Ga-NOTA-T4 or [18F]AlF-RESCA-T4 will help select patients for targeted therapy and monitor treatment responses after the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Be between 18 and 65 years of age and of either sex.
2. Patients with colorectal cancer confirmed by puncture or surgical pathology.
3. Written informed consent signed by the subject or legal guardian or caregiver.
4. Willingness and ability to cooperate with all programs of this study.

Exclusion Criteria:

1. Severe hepatic or renal insufficiency;
2. Targeted therapy before radiotherapy or PET/CT scan；
3. Renal function: serum creatinine less than or equal to the upper limit of the normal range;Liver function: bilirubin, AST(SGOT)/ALT(SGPT) less than or equal to the upper limit of the normal range；
4. History of serious surgery in the last month. Those who have participated in other clinical trials during the same period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
evaluate the safety and feasibility of [68Ga]Ga-NOTA-T4 or [18F]AlF-RESCA-T4 PET/CT imaging in patients with solid tumors | 1 hour after injection of [68Ga]Ga-NOTA-T4 or [18F]AlF-RESCA-T4
  The primary goal of the study is to evaluate the distribution profiles (in terms of SUVmax) of [68Ga]Ga-NOTA-T4 or [18F]AlF-RESCA-T4 PET/CT imaging in patients with solid tumors.
evaluate the sensitivity and specificity of [68Ga]Ga-NOTA-T4 or [18F]AlF-RESCA-T4 PET/CT for visualizing TROP-2 expression | 1 hour after injection of [68Ga]Ga-NOTA-T4 or [18F]AlF-RESCA-T4
  The secondary goal is to evaluate the sensitivity and specificity of [68Ga]Ga-NOTA-T4 or [18F]AlF-RESCA-T4 PET/CT for visualizing TROP-2 expression.
evaluate the value of TROP-2 expression determined by [68Ga]Ga-NOTA-T4 or [18F]AlF-RESCA-T4 PET/CT | 1 hour after injection of [68Ga]Ga-NOTA-T4 or [18F]AlF-RESCA-T4
  The third goal is to evaluate the value of TROP-2 expression determined by [68Ga]Ga-NOTA-T4 or [18F]AlF-RESCA-T4 PET/CT in differential diagnosis, patient selection, and response monitoring in patients with solid tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Xie, PhD, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, China